CLINICAL TRIAL: NCT06727318
Title: Comparison of Capillary Refill Time and Serum Lactate Level in Predicting Disease Prognosis in Patients With Septic Shock
Brief Title: Comparison of Peripheral Perfusion Indicators and Lactate Levels
Status: Completed | Type: Observational
Sponsor: Gulhane Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Mete Erdemir, İNTENSİVE CARE SPECİALİST, Gulhane Training and Research Hospital
Other Study IDs: 2024/208
Record Dates: First submitted 2024-11-15; First posted 2024-12-10 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2024-05

CONDITIONS: Sepsis; Shock, Septic; Hypotensive; Lactate; Lactic Acidosis
Keywords: SEPSİS; SEPTİC SHOCK; CAPİLLER REFİLL TİME; LACTATE İNCRASE; HYPOTENSİVE
MeSH Terms: conditions — Sepsis; Shock, Septic; Acidosis, Lactic; Toxemia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In patients with septic shock undergoing intensive care unit monitoring, routine assessment of arterial and/or venous blood gas is conducted. During the period when arterial and/or venous blood gas is analyzed in this patient cohort, peripheral perfusion indicators will also be examined. Peripheral perfusion indicators will be appraised using capillary refill and mottling score. In patients experiencing septic shock, elevated lactate levels and progressive elevation of lactate levels during monitoring, prolonged capillary refill time exceeding 3 seconds, protracted capillary refill time, mottling development, and escalating mottling score are prognostic indicators of poor outcomes. The objective of this prospective study is to assess the correlation between capillary refill time and mottling score, concurrently evaluated, and serum lactate levels in arterial and/or venous blood gas.

DETAILED DESCRIPTION:
Sepsis is defined as life-threatening organ dysfunction caused by dysregulated host response to infection(1). Patients with septic shock can be characterized by a clinical table of sepsis with a serum lactate level >2 mmol/L (18mg/dL) despite adequate fluid resuscitation and persistent hypotension requiring vasopressors to maintain a mean arterial pressure (MAP) ≥65 mm Hg (2). Shock is characterized by signs of tissue hypoperfusion, including increased serum lactate levels and abnormal peripheral perfusion (3). Mottling of the leg is a finding indicating impaired peripheral perfusion(4). Inadequate reduction of high lactate levels with treatment has been associated with an increased risk of death(5). Demographic data of all patients (age, gender, educational status, occupation), comorbidities, APACHE-II score, SOFA score, Charlson Comorbidity index, SAPS-II, MV support, service of transfer to intensive care unit, day of septic shock diagnosis; CRP, procalcitonin, albumin, fibrinogen, WBC, neutrophil count, lymphocyte, platelet count, INR, culture results, disseminated intravascular coagulation (DIC) score, capillary refill, mottling score, blood gas serum lactate level and base deficit, arterial pCO2 value, venous pCO2 value, arterio-venous PCO2 gradient difference, urine volume, vasopressor dose, mean arterial pressure and other vital signs will be noted. Arterial and/or venous blood gases measured every 6 hours from the time of diagnosis and concurrent peripheral perfusion findings (capillary refill time, mottling score) will be noted in the first 24 hours. Capillary refill time was planned to be measured by applying strong pressure to the ventral surface of the distal phalanx of the right index finger with a glass microscope slide. The pressure was planned to continue for 10 seconds after the nail bed turned white. The time to return to normal skin color will be recorded with a chronometer and a refill time longer than 3 seconds will be considered abnormal. In addition, mottling score will be examined as another peripheral perfusion examination outcome. Mottling score is as described below; If there is no mottling, the score will be considered as 0. If there is a coin-sized mottled discoloration in the knee, the score will be evaluated as 1, if the discoloration continues to the upper part of the kneecap, the score will be evaluated as 2, if it reaches to the middle of the thigh, the score will be evaluated as 3, if it reaches to the groin, the score will be evaluated as 4, and if the discoloration exceeds the groin area, the score will be evaluated as 5. Thus, blood gas and peripheral perfusion findings will be noted every 6 hours in the first 24 hours after the patients who are followed up in the intensive care unit with a diagnosis of septic shock and who meet the inclusion criteria are included in the study.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Patients in septic shock

Exclusion Criteria:

* Patients who did not give consent for participation in the study
* Patients under 18 years of age
* Patients with aortic pathology
* Patients with arrhythmias (arrhythmias affecting cardiac index)
* Patients with peripheral arterial disease (Buerger's disease, etc.)
* Patients with a diagnosis of Raynaud's disease
* Patients with chronic liver disease
* Black people
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Septic shock patients in the intensive care unit
Sampling Method: Non-Probability Sample
Enrollment: 192 (Actual)
Dates: Start 2024-05-01 (Actual); Primary Completion 2025-08-18 (Actual); Study Completion 2025-08-18 (Actual)

PRIMARY OUTCOMES:
USE OF PERİFERAL PERFUSİON ASSESSMENT METHODS | MAY 2024 SEPTEMBER 2025
  Arterial and/or venous blood gases measured every 6 hours from the time of diagnosis and concurrent peripheral perfusion findings (capillary refill time, mottling score) will be noted in the first 24 hours. Capillary refill time, mottling score, lactate level measurements will be evaluated separately for septic shock progression and 28-day mortality. Parameters that are significant for septic shock progression in univariate analysis will be evaluated with logistic regression analysis. Then, the correlation between the peripheral perfusion findings and lactate levels will be compared with correlation analysis.

CONTACTS AND LOCATIONS:
Locations (1):
- Healty Sciences University Gulhane Training and Research Hospital, Ankara, KEÇİÖREN, Turkey (Türkiye)

REFERENCES:
- [Result] Stevenson LW, Perloff JK. The limited reliability of physical signs for estimating hemodynamics in chronic heart failure. JAMA. 1989 Feb 10;261(6):884-8. PMID 2913385
- [Result] Ait-Oufella H, Lemoinne S, Boelle PY, Galbois A, Baudel JL, Lemant J, Joffre J, Margetis D, Guidet B, Maury E, Offenstadt G. Mottling score predicts survival in septic shock. Intensive Care Med. 2011 May;37(5):801-7. doi: 10.1007/s00134-011-2163-y. Epub 2011 Mar 4. PMID 21373821
- [Result] Cecconi M, De Backer D, Antonelli M, Beale R, Bakker J, Hofer C, Jaeschke R, Mebazaa A, Pinsky MR, Teboul JL, Vincent JL, Rhodes A. Consensus on circulatory shock and hemodynamic monitoring. Task force of the European Society of Intensive Care Medicine. Intensive Care Med. 2014 Dec;40(12):1795-815. doi: 10.1007/s00134-014-3525-z. Epub 2014 Nov 13. PMID 25392034
- [Result] Singer M, Deutschman CS, Seymour CW, Shankar-Hari M, Annane D, Bauer M, Bellomo R, Bernard GR, Chiche JD, Coopersmith CM, Hotchkiss RS, Levy MM, Marshall JC, Martin GS, Opal SM, Rubenfeld GD, van der Poll T, Vincent JL, Angus DC. The Third International Consensus Definitions for Sepsis and Septic Shock (Sepsis-3). JAMA. 2016 Feb 23;315(8):801-10. doi: 10.1001/jama.2016.0287. PMID 26903338